CLINICAL TRIAL: NCT02324361
Title: Quincy Family, Youth & Technology For Lifestyle Change (FYT-4-LIFE) Study
Acronym: QFYT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000873
Record Dates: First submitted 2014-07-07; First posted 2014-12-24 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Obesity
Keywords: Pediatric; Obesity; Intervention; Information and Communication Technologies; Social Media; Text Messaging; Mobile Health
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2-arm interventional study
Masking Description: Participants were given a choice to select one of the two interventions, which were made clear to them. There was no masking of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook group (Experimental): The intervention consists of evidence-based information on healthy family routines and parenting strategies adapted for Facebook posts on a private study Facebook group.
  Participating parents/guardians will have access to all features of the secret study Facebook group (e.g., create and view postings, comment and like existing posts and view user names of other members of the group (existing study participants and staff) for the duration of the study.
  All index children will be provided with a Physical Activity Monitor to wear during waking hours for the duration of the study.
  Interventions: Other: Physical Activity; Behavioral: Evidence-based information on healthy family routines
- Text messaging (Experimental): The intervention consists of evidence-based information on healthy family routines and parenting strategies adapted for 140-character text messages.
  The automated text-messaging algorithm consists of the delivery of two types of text messages: 1-way messages, in which participating parents/guardians will receive a piece of education or motivation on the dimension topic that they're being coached on and 2-way messages, in which participants are able to respond to an educational message containing a number response prompt that will provide them with personalized feedback regarding a dimension they are being coached on.
  All index children will be provided with a Physical Activity Monitor to wear during waking hours for the duration of the study.
  Interventions: Other: Physical Activity; Behavioral: Evidence-based information on healthy family routines

INTERVENTIONS:
Other: Physical Activity — The Fitbit Zip is a wireless physical activity monitor that will be worn by the index child during waking hours, and will be used to assess daily active time for the duration of the study.
  Other Names: Change in Physical Activity
Behavioral: Evidence-based information on healthy family routines — Educational dimensions include nutrition, frequency of family meals, child's screen time, bedtime routines, physical activity, and sleep hours.

SUMMARY:
To date, approaches that show the most promise for preventing and/or reversing the course of childhood obesity involve the delivery of intensive lifestyle interventions within a family-based context, emphasizing the necessity of parental involvement and making changes in family routines and the home environment. Considering that the current demand for pediatric weight management programs far exceed availability, as well as the high attrition rates observed in such programs, there is a great need for more accessible and efficient means of delivering these interventions to reduce the burden of childhood obesity.

The goal of this study is to understand whether text messaging and social media platforms can be leveraged to address the important issue of childhood obesity by engaging parent/guardians in one of these strategies, and whether these strategies produce similar outcomes. No existing study has compared these strategies head-to-head, and the investigators believe that this project will be instrumental in understanding the determinants of success in these strategies and allow us to collect sufficient intelligence to be able to deploy these meaningfully to patients as part of usual care.

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate and compare the feasibility and effectiveness of two platforms, text messaging and Facebook, for delivering an evidence-based, family-centric childhood obesity intervention to parent/guardians of children between the ages of 3-6 with a BMI of 90th percentile and above. The investigators hypothesize that the use of both platforms for delivering a childhood obesity intervention will help establish healthier family routines and be equally engaging and accepted by parent/guardians and children.

The primary aim of this study is to assess the effect of the intervention on:

* Parent/guardian knowledge of healthy family routines (i.e., nutrition, frequency of family meals, child's screen time, bedtime routines, physical activity, and sleep hours) and of parenting strategies that are preventive of child overweight and obesity
* Parent/guardian readiness, confidence, and perceived self-efficacy to make and maintain changes in family routines known to be associated with healthy weight outcomes

The secondary aims of the study are to assess the effect of the intervention on:

* The adoption of healthy family routines and parenting strategies that are preventive of child overweight and obesity
* Daily objective physical activity in the index child by accelerometry (using a physical activity tracking device)
* Index children's BMI percentile, using data collected during regular clinic visits from the electronic medical record
* To assess the level of engagement with the intervention, measured via daily activity tracker wear by the index child, parent/guardian views of Facebook posts or responses to 2-way text messages

ELIGIBILITY:
Inclusion Criteria:

* Index child's BMI ≥90th percentile
* Index child age between 3 and 7 years of age at time of enrollment in study
* The child is under the care of a primary care provider at the Quincy Pediatric Associates practice
* The family is not planning to move from the Greater Boston area during the study period

The participating parent/guardian:

* Is 18 years or older
* Is the primary caregiver for the child
* Has regular access to the Internet
* Has regular access to a personal computer with USB connection OR a smartphone with a mobile operating system that is compatible with the physical activity tracker
* Owns a Facebook account AND a cellphone with text messaging capability and if choosing the text-messaging intervention, is willing to receive a maximum of 62 text messages/month for 3 months on their personal cellphone
* Is fluent in English (spoken and written)

Exclusion Criteria:

* Children who are diagnosed with underlying medical or pharmacologic factors that may contribute to obesity and/or affect participation in physical activity
* Significant medical or psychiatric co-morbidities in the participating parent/guardian
* Visual, hearing, or cognitive impairments in the participating parent/guardian
* Index child or parent/guardian currently enrolled in another weight control program
* Children who have a sibling already enrolled in the study

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Quincy Pediatric Associates, Quincy, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July to October 2014, attempts were made to solicit the participation of primary caregivers of all children receiving care since 2013 at Quincy Pediatric Associates (QPA) via mailed recruitment letters.
Pre-assignment Details: Caregivers were phone-screened for English fluency, internet access, computer/smartphone ownership, and ownership of a Facebook account. Those with significant functional impairments or co-morbidities, those enrolled in another weight management intervention program, or had a sibling already enrolled in the study were excluded from participation.
Groups:
- Facebook Group: The intervention arm consists of evidence-based information on healthy family routines and parenting strategies (i.e., nutrition, frequency of family meals, child's screen time, bedtime routines, physical activity, and sleep) adapted for Facebook posts on a private study Facebook group.
  All index children were provided with a Physical Activity Monitor (Fitbit Zip) to wear during waking hours for the duration of the study.
- Text Messaging (SMS) Group: The intervention consists of evidence-based information on healthy family routines and parenting strategies adapted for 140-character text messages.
  The automated text-messaging algorithm consists two types of messaging: 1-way messages containing education or motivation on the dimension topic that one is being coached on and 2-way messages, in which participants are able to respond to an educational message containing a number response prompt that will provide them with personalized feedback regarding a dimension they are being coached on.
  All index children were provided with a Physical Activity Monitor (Fitbit Zip) to wear during waking hours for the duration of the study.
Period: Overall Study
Arm/Group | Facebook Group | Text Messaging (SMS) Group
Started | 24 | 24
Completed | 19 | 22
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: 1 participant from the Facebook group was unresponsive to contact and subsequently omitted from baseline analysis.
Groups:
- Text Messaging: The intervention consists of evidence-based information on healthy family routines and parenting strategies adapted for 140-character text messages.
  The automated text-messaging algorithm consists of the delivery of two types of text messages: 1-way messages, in which participating parents/guardians will receive a piece of education or motivation on the dimension topic that they're being coached on and 2-way messages, in which participants are able to respond to an educational message containing a number response prompt that will provide them with personalized feedback regarding a dimension they are being coached on.
- Total: Total of all reporting groups
Arm/Group | Facebook Group | Text Messaging | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of caregiver
  years | 38.4 (5.3) | 40.2 (9.9) | 39.3 (7.9)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of index child
  years | 4.9 (1.3) | 5.3 (1.3) | 5.0 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of index child
  Participants
    Female | 9 | 14 | 23
    Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver ethnicity
  Participants
    Hispanic or Latino | 0 | 3 | 3
    Not Hispanic or Latino | 23 | 21 | 44
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 4 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 21 | 19 | 40
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Parent/Guardian Knowledge of Healthy Family Routines and of Parenting Strategies That Are Preventive of Child Overweight and Obesity
Description: We designed a scale for use in this study containing 8 questions on each of the family routines that we assessed (i.e., nutrition, frequency of family meals, child's screen time, bedtime routines, physical activity, and sleep hours). Each of the eight questions were assigned one point value. The scale was summative such that the lowest possible score was 0 and highest possible score was 8, from adding up scores to all eight questions. Higher scores indicated a better outcome.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Facebook Group | Text Messaging (SMS) Group
Number analyzed (Participants) | 23 | 24
units on a scale | 1.2 [0.6 to 1.7] | 0.9 [0.2 to 1.6]

2. Secondary Outcome: Change in Sleep
Description: Baseline to 90-days post-intervention change in child sleep duration (hours per day)
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: hours per day
Arm/Group | Facebook Group | Text Messaging (SMS) Group
Number analyzed (Participants) | 23 | 24
hours per day | 0.3 [-0.8 to 0.7] | 0.3 [0.0 to 0.5]

3. Secondary Outcome: Change in Child Screen Time Exposure
Description: Baseline to 90-days post-intervention change in child screen time exposure (hours per day)
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: hours per day
Arm/Group | Facebook Group | Text Messaging (SMS) Group
Number analyzed (Participants) | 23 | 24
hours per day | -0.7 [-1.5 to 0.1] | -0.4 [-1.1 to 0.4]

4. Secondary Outcome: Change in Sugar Sweetened Beverage Intake
Description: Baseline to 90-days post-intervention change in child sugar sweetened beverage intake (servings per day)
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: servings per day
Arm/Group | Facebook Group | Text Messaging (SMS) Group
Number analyzed (Participants) | 23 | 24
servings per day | -0.1 [-0.3 to 0.2] | -0.4 [-0.8 to 0.0]

ADVERSE EVENTS:
Time Frame: 90 days, over the entire duration of the study
Arm/Group | Facebook Group | Text Messaging (SMS) Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

LIMITATIONS AND CAVEATS:
Having participants self-select the technology platform used to deliver an mHealth intervention may promote intervention engagement this lack of randomization potentially limits the generalizability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No